CLINICAL TRIAL: NCT02392780
Title: Cannabidiol for the Treatment of Severe (Grades III/IV) Acute Graft-versus-host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: moshe yeshurun (Other)
Responsible Party: Sponsor-Investigator, moshe yeshurun, Head, BMT unit, Rabin Medical Center, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0009-15-RMC
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Acute-graft-versus-host Disease
MeSH Terms: interventions — Cannabidiol; Methylprednisolone; Calcineurin Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cannabidiol (Experimental)
  Interventions: Drug: Cannabidiol; Drug: Methylprednisolone; Drug: Calcineurin inhibitor

INTERVENTIONS:
Drug: Cannabidiol — Oral cannabidiol at a dose of 150 mg BID up to 90 days.
Drug: Methylprednisolone — IV methylprednisolone 2 mg/kg/day
Drug: Calcineurin inhibitor — cyclosporine with dose adjusted based on drug trough levels (200-400 ng/ml) or tacrolimus with dose adjusted on drug trough levels (5-15 ng/ml)

SUMMARY:
Graft-versus-host-disease (GVHD) is a major obstacle to successful allogeneic hematopoietic cell transplantation (alloHCT). Cannabidiol (CBD), a non-psychotropic ingredient of Cannabis sativa possesses potent anti-inflammatory and immunosuppressive properties. In a recent phase 2 study, CBD has been shown to be safe and reduced significantly the incidence of acute GVHD compared to control patients with a hazard ratio of 0.3. Based on these results the investigators propose a phase 2 study to explore the efficacy of oral CBD in the treatment of severe (grades III/IV) acute GVHD, a pathology with a dismal prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. After allogeneic transplantation
3. Grade III or IV acute GVHD
4. No psychiatric contra-indication
5. Informed consent

Exclusion Criteria:

1. History of psychosis
2. Asthma
3. Known allergy to cannabis constituents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete remission of acute GVHD | 90 days

SECONDARY OUTCOMES:
Proportion of patients with partial remission of acute GVHD | 90 days
Proportion of patients with chronic GVHD | 12 months
Proportion of patients able to discontinue immunosuppression | 12 months
Transplant related mortality | 12 months

OTHER OUTCOMES:
Subpopulations of peripheral blood cells and cytokine levels | 12 months
  T4, T8, Foxp3 T regulatory cells, TNFα, INFγ, IL-1β, IL-6, IL-17, IL-4, IL-5, IL-10 and IL-13

CONTACTS AND LOCATIONS:
Locations (1):
- Davidof Cancer Center, Beilinson hospital, Rabin medical center, Petah Tikva, Israel